CLINICAL TRIAL: NCT05920655
Title: Comparison of Ocular Changes by Surgical Menopause Using Optical Coherence Tomography (OCT)
Status: Completed | Type: Observational
Sponsor: Batman Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erhan Okuyan,M.D, M.D, Batman Training and Research Hospital
Other Study IDs: 2023
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Corneal Deformity; Macular Degeneration Advanced; Surgical Menopause

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1( Surgical menopause): Surgical menopause : At least 6 months after hysterectomy and salphingo-oopherectomy
  Interventions: Diagnostic Test: Optic coherence tomography
- 2 ( Natural menopause ): Natural menopause :Healthy female patients who have not had a menstrual period for at least 1 year and have not received any treatment for this reason before
  Interventions: Diagnostic Test: Optic coherence tomography
- 3 (Control ): Healthy women aged 30-45 years with regular menstrual cycles and no symptoms of menopause
  Interventions: Diagnostic Test: Optic coherence tomography

INTERVENTIONS:
Diagnostic Test: Optic coherence tomography — Eye examination of patients with optic coherence tomography test by an ophthalmologist

SUMMARY:
The aim of this study is to investigate the early changes in macular thickness, corneal thickness and intraocular pressure in young women undergoing surgical menopause.

Methods: Eye findings of 30 surgical menopausal (Postoperative 3-6 months) and 48 natural menopause and 22 healty women (control) were evaluated using OCT. Women with no known eye disease, no chronic disease (Diabetes Mellitus, Cardiac Disease any Autoimmune disease) and no migraine in addition to non smokers were included in the study. Women using any hormone and obese women ( BMI >25 kg/m2) were excluded. Macular and corneal thickness and intraocular pressure (IOP) were measured in both eyes of the women

DETAILED DESCRIPTION:
This prospective case control study was conducted in a tertiary gynecology and obstetrics clinic and eye clinic between 2020 and 2021 with ethics committee approval number 2020 250 ). Informed consent form was obtained from all participants. All participants were outpatients who applied to obstetrics clinic in Batman Training and Research Hospital.

The study started with 105 patient. Based on the study exclusion criteria, 7 patients were excluded from the study. Every patient in the surgical menopause group underwent a hysterectomy and bilateral salpingo-oophorectomy for benign uterine reasons. The patients included in the study were menstruating women with preoperative natural ovarian appearance and benign non ovarian indications, who had undergone hysterectomy and bilateral salpingo-oophorectomy and had no preoperative menopause complaints. Patients younger than 52 years of age who have undergone oophorectomy are patients whose ovaries have been removed either because of patient anxiety due to a family history of cancer or because of adhesions.

ELIGIBILITY:
Inclusion Criteria:

* The patients included in the study were menstruating women with preoperative natural ovarian appearance and benign non ovarian indications, who had undergone hysterectomy and bilateral salpingo-oopherectomy, and had no preoperative menopause complaints. Patients younger than 52 years of age who have undergone oophorectomy are patients whose ovaries have been removed either because of patient anxiety due to a family history of cancer or because of adhesions.
* having a healthy child
* have consented to participate in the study

Exclusion Criteria:

* Chronic disease (such as diabetes, heart disease)
* History of continuous drug use
* Unwillingness to participate in the study Being between the ages of 18-30

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female ,age between 30-55 .
Study Population: Patient selection was made between surgical menopause, natural menopause and healthy women who have given birth before.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Effect of surgical menopause on corneal and macular thickness | 6 months after hysterectomy and bilateral salpingo-oopherectomy
  To question the effect on macular and corneal thickness secondary to sudden ovarian hormone change with surgical menopause.

SECONDARY OUTCOMES:
Eye examination needed after surgical menopause | 6-12 months
  To seek an answer to the question of adding eye diseases examination to the examinations of post-surgical menopause patients.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Okuyan, Principal Investigator — Batman Training and Research Hospital
Locations (1):
- Batman education adn research hospital, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Will be given to the journal upon request.